CLINICAL TRIAL: NCT03867058
Title: Tradeoff Between Spatial Resolution of Neural Excitation and Temporal Rate Processing
Brief Title: Tradeoff Between Spatial and Temporal Resolution
Status: Terminated | Type: Observational
Why Stopped: PI passed away. Ending grant and closing lab.
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Heather Wright, professor, East Carolina University
Other Study IDs: Zhou_R01_study1
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cochlear implant users with Nucleus and AB devices: Temporal processing acuity will be compared using electrodes or electrode configurations that create broad versus sharp spatial excitation.
  Speech recognition will be compared in the same group of subjects using electrode-dependent focused versus monopolar stimulation.
  Interventions: Behavioral: Electrode selection/electrode configuration

INTERVENTIONS:
Behavioral: Electrode selection/electrode configuration — Electrodes will be chosen based on their spatial tuning curves. Focused stimulation will be applied to electrodes with good temporal processing acuity.

SUMMARY:
In this study, investigators will examine how temporal rate processing might be affected when the width of neural excitation narrows. The manipulation of neural excitation width will be achieved for example by changing electrode configurations or stimulating single versus multiple electrodes simultaneously. Investigators will then measure if the extent to which rate processing is affected by spatially restricted stimulation can predict a subject's overall speech recognition and predict also whether the subject is likely to benefit from a focused electrode configuration. Lastly, investigators will introduce and test a novel current focusing strategy where current focusing is applied in a channel specific manner and quantify if this intervention improves speech recognition. The primary endpoint of the study is speech recognition, and the secondary endpoint is psychophysical sensitivity to stimulation rate change.

ELIGIBILITY:
Inclusion Criteria:

* Native speakers of English
* Cochlear Nucleus cochlear implant users or Advanced Bionics users
* Postlingually deafened
* Has had device experience for at least one year
* Can be child or adult at the time of enrollment

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults received cochlear implants (Advanced Bionics and Cochlear Nucleus devices).
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Sensitivity to stimulation rate change at threshold | starting 6 months post award notice and will take up to 4 years to complete
  Subjects' psychophysical detection thresholds will be measured as a function of the rate of stimulation delivered to selected electrodes and selected electrode configuration
Discrimination of stimulation rate | starting 6 months post award notice and will take up to 4 years to complete
  subjects' ability to discriminate stimulation rates will be measured as a function of base stimulation rates at selected electrodes and selected electrode configuration.

SECONDARY OUTCOMES:
Speech recognition | starting 6 months post award notice and will take up to 4 years to complete
  Speech recognition in quiet and in noise will be measured under three conditions: 1. the traditional monopolar electrode configuration; 2. using current focusing on electrodes that show good sensitivity to rate change; 3. using current focusing on all electrodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Communication Sciences and Disorders, ECU, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chatterjee M, Galvin JJ 3rd, Fu QJ, Shannon RV. Effects of stimulation mode, level and location on forward-masked excitation patterns in cochlear implant patients. J Assoc Res Otolaryngol. 2006 Mar;7(1):15-25. doi: 10.1007/s10162-005-0019-2. Epub 2005 Nov 4. PMID 16270234
- [Background] Nelson DA, Kreft HA, Anderson ES, Donaldson GS. Spatial tuning curves from apical, middle, and basal electrodes in cochlear implant users. J Acoust Soc Am. 2011 Jun;129(6):3916-33. doi: 10.1121/1.3583503. PMID 21682414
- [Background] Bierer JA, Litvak L. Reducing Channel Interaction Through Cochlear Implant Programming May Improve Speech Perception: Current Focusing and Channel Deactivation. Trends Hear. 2016 Jun 17;20:2331216516653389. doi: 10.1177/2331216516653389. PMID 27317668
- [Background] Berenstein CK, Mens LH, Mulder JJ, Vanpoucke FJ. Current steering and current focusing in cochlear implants: comparison of monopolar, tripolar, and virtual channel electrode configurations. Ear Hear. 2008 Apr;29(2):250-60. doi: 10.1097/aud.0b013e3181645336. PMID 18595189
- [Background] Boulet J, White M, Bruce IC. Temporal Considerations for Stimulating Spiral Ganglion Neurons with Cochlear Implants. J Assoc Res Otolaryngol. 2016 Feb;17(1):1-17. doi: 10.1007/s10162-015-0545-5. PMID 26501873
- [Background] Carlyon RP, Deeks JM. Combined neural and behavioural measures of temporal pitch perception in cochlear implant users. J Acoust Soc Am. 2015 Nov;138(5):2885-905. doi: 10.1121/1.4934275. PMID 26627764
- [Background] Carlyon RP, Deeks JM. Limitations on rate discrimination. J Acoust Soc Am. 2002 Sep;112(3 Pt 1):1009-25. doi: 10.1121/1.1496766. PMID 12243150
- [Background] Dingemanse JG, Frijns JH, Briaire JJ. Psychophysical assessment of spatial spread of excitation in electrical hearing with single and dual electrode contact maskers. Ear Hear. 2006 Dec;27(6):645-57. doi: 10.1097/01.aud.0000246683.29611.1b. PMID 17086076
- [Background] Eggermont JJ. Peripheral auditory adaptation and fatigue: a model oriented review. Hear Res. 1985 Apr;18(1):57-71. doi: 10.1016/0378-5955(85)90110-8. PMID 2993220
- [Background] Galvin JJ 3rd, Fu QJ. Effects of stimulation rate, mode and level on modulation detection by cochlear implant users. J Assoc Res Otolaryngol. 2005 Sep;6(3):269-79. doi: 10.1007/s10162-005-0007-6. PMID 16075190
- [Background] Green T, Faulkner A, Rosen S. Variations in carrier pulse rate and the perception of amplitude modulation in cochlear implant users. Ear Hear. 2012 Mar-Apr;33(2):221-30. doi: 10.1097/AUD.0b013e318230fff8. PMID 22367093
- [Background] Goldsworthy RL, Shannon RV. Training improves cochlear implant rate discrimination on a psychophysical task. J Acoust Soc Am. 2014 Jan;135(1):334-41. doi: 10.1121/1.4835735. PMID 24437773
- [Background] Javel E, Shepherd RK. Electrical stimulation of the auditory nerve. III. Response initiation sites and temporal fine structure. Hear Res. 2000 Feb;140(1-2):45-76. doi: 10.1016/s0378-5955(99)00186-0. PMID 10675635
- [Background] Kreft HA, Oxenham AJ, Nelson DA. Modulation rate discrimination using half-wave rectified and sinusoidally amplitude modulated stimuli in cochlear-implant users. J Acoust Soc Am. 2010 Feb;127(2):656-9. doi: 10.1121/1.3282947. PMID 20136187
- [Background] Kwon BJ, van den Honert C. Effect of electrode configuration on psychophysical forward masking in cochlear implant listeners. J Acoust Soc Am. 2006 May;119(5 Pt 1):2994-3002. doi: 10.1121/1.2184128. PMID 16708955
- [Background] Landsberger DM. Effects of modulation wave shape on modulation frequency discrimination with electrical hearing. J Acoust Soc Am. 2008 Aug;124(2):EL21-7. doi: 10.1121/1.2947624. PMID 18681497
- [Background] Macherey O, Carlyon RP. Re-examining the upper limit of temporal pitch. J Acoust Soc Am. 2014 Dec;136(6):3186. doi: 10.1121/1.4900917. PMID 25480066
- [Background] McDermott HJ, McKay CM. Musical pitch perception with electrical stimulation of the cochlea. J Acoust Soc Am. 1997 Mar;101(3):1622-31. doi: 10.1121/1.418177. PMID 9069629
- [Background] McKay CM, McDermott HJ. Loudness perception with pulsatile electrical stimulation: the effect of interpulse intervals. J Acoust Soc Am. 1998 Aug;104(2 Pt 1):1061-74. doi: 10.1121/1.423316. PMID 9714925
- [Background] Miller CA, Woo J, Abbas PJ, Hu N, Robinson BK. Neural masking by sub-threshold electric stimuli: animal and computer model results. J Assoc Res Otolaryngol. 2011 Apr;12(2):219-32. doi: 10.1007/s10162-010-0249-9. Epub 2010 Nov 16. PMID 21080206
- [Background] Moore BC. Frequency difference limens for short-duration tones. J Acoust Soc Am. 1973 Sep;54(3):610-9. doi: 10.1121/1.1913640. No abstract available. PMID 4754385
- [Background] Nilsson M, Soli SD, Sullivan JA. Development of the Hearing in Noise Test for the measurement of speech reception thresholds in quiet and in noise. J Acoust Soc Am. 1994 Feb;95(2):1085-99. doi: 10.1121/1.408469. PMID 8132902
- [Background] Pijl S, Schwarz DW. Melody recognition and musical interval perception by deaf subjects stimulated with electrical pulse trains through single cochlear implant electrodes. J Acoust Soc Am. 1995 Aug;98(2 Pt 1):886-95. doi: 10.1121/1.413514. PMID 7642827
- [Background] Thornton AR, Raffin MJ. Speech-discrimination scores modeled as a binomial variable. J Speech Hear Res. 1978 Sep;21(3):507-18. doi: 10.1044/jshr.2103.507. PMID 713519